CLINICAL TRIAL: NCT06818643
Title: A Phase 1/2 Open-label Study to Evaluate the Safety and Efficacy of MK-3120 in Participants With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Efficacy of MK-3120 in Participants With Advanced Solid Tumors (MK-3120-002)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3120-002; 2024-516817-19-00 (Registry Identifier: EU CT); U1111-1311-1904 (Registry Identifier: UTN); jRCT2031250198 (Registry Identifier: Japan Registry of Clinical Trial (jRCT))
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Dose level 1 (Experimental): Participants receive MK-3120 at dose level 1 as per the schedule specified in the arm.
  Interventions: Biological: MK-3120
- Arm 2 Dose level 2 (Experimental): Participants receive MK-3120 at dose level 2 as per the schedule specified in the arm.
  Interventions: Biological: MK-3120

INTERVENTIONS:
Biological: MK-3120 — IV infusion
  Other Names: SKB410

SUMMARY:
Researchers are looking for new ways to treat people with certain advanced solid tumors. Advanced means the cancer has spread to other parts of the body and cannot be removed with surgery. Solid tumors are cancers mostly in body organs and tissues, not in the blood or other body liquids. The main goal of this study is to learn about the safety of MK-3120 and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed advanced (unresectable and/or metastatic) solid tumor and has received or been intolerant to all available treatments
* If human immunodeficiency virus (HIV) positive, has well controlled HIV on antiretroviral therapy (ART)
* If hepatitis B surface antigen (HBsAg) positive, must have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load
* If hepatitis C virus (HCV) infected, must have undetectable HCV viral load

Exclusion Criteria:

* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled significant cardiovascular disease or cerebrovascular disease
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has pleural effusion, ascites, and/or pericardial effusion that are symptomatic or require repeated drainage
* Is HIV-positive and has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Known additional malignancy that is progressing or has required active treatment within the past 2 years
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active infection requiring systemic therapy, with exceptions
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has HBV or HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-10-25 (Estimated); Study Completion 2031-03-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 43 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 42 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) as Assessed by the Investigator | Up to approximately 72 months
  ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by the investigator per RECIST 1.1.
Duration Of Response (DOR) Per RECIST 1.1 as Assessed by the Investigator | Up to approximately 72 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by the investigator per RECIST 1.1 will be presented.
Progression-free Survival (PFS) Per RECIST 1.1 as Assessed by the Investigator | Up to approximately 72 months
  PFS is defined as the time from the first dose of study treatment to the first documented PD or death due to any cause, whichever occurs first will be assessed by the investigator using RECIST 1.1. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by the investigator per RECIST 1.1 will be presented.
Overall Survival (OS) Per RECIST 1.1 as Assessed by the Investigator | Up to approximately 72 months
  OS is defined as the time from the first dose of study treatment to death due to any cause as assessed by the investigator per RECIST 1.1 will be presented.
Area Under the Concentration-Time Curve (AUC) of MK-3120 Antibody-Drug Conjugate (ADC) | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the AUC of MK-3120 ADC.
AUC of MK-3120 Total Antibody (TAb) | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the AUC of MK-3120 TAb
AUC of MK-3120 Free Payload | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the AUC of MK-3120 free payload.
Maximum Concentration (Cmax) of MK-3120 ADC | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmax of MK-3120 ADC.
Cmax of MK-3120 TAb | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmax of MK-3120 TAb.
Cmax of MK-3120 Free Payload | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmax of MK-3120 free payload.
Minimum Concentration (Cmin) of MK-3120 ADC | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmin of MK-3120 ADC.
Cmin of MK-3120 TAb | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmin of MK-3120 TAb.
Cmin of MK-3120 Free Payload | At specified time points up to approximately 43 months
  Blood samples will be collected to determine the Cmin of MK-3120 free payload.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (42):
- United States (4):
  - The University of Alabama at Birmingham ( Site 1005), Birmingham, Alabama
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 1003), Miami, Florida
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1009), Hackensack, New Jersey
  - Virginia Commonwealth University ( Site 1008), Richmond, Virginia
- Chile (4):
  - Centro de Estudios Clínicos SAGA ( Site 0033), Santiago, Region M. de Santiago
  - FALP ( Site 0031), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0032), Santiago, Region M. de Santiago
  - Bradford Hill Centro de Investigaciones Clinicas ( Site 0030), Santiago, Region M. de Santiago
- China (5):
  - Peking University First Hospital ( Site 0180), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 0186), Chongqing, Chongqing Municipality
  - Hunan Cancer Hospital ( Site 0181), Changsha, Hunan
  - The First Hospital of Jilin University ( Site 0185), Changchun, Jilin
  - West China Hospital Sichuan University ( Site 0187), Chengdu, Sichuan
- France (4):
  - Institut Paoli Calmettes ( Site 0053), Marseille, Bouches-du-Rhone
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer-Medical Oncology ( Site 0054), Rennes, Ille-et-Vilaine
  - Centre Oscar Lambret ( Site 0051), Lille, Nord
  - Gustave Roussy ( Site 0050), Villejuif, Val-de-Marne
- Israel (3):
  - Rambam Health Care Campus ( Site 0082), Haifa
  - Rabin Medical Center ( Site 0081), Petah Tikva
  - Sheba Medical Center ( Site 0080), Ramat Gan
- Japan (3):
  - National Cancer Center Hospital East ( Site 0190), Kashiwa, Chiba
  - Cancer Institute Hospital of JFCR ( Site 0192), Koto, Tokyo
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 0191), Osaka
- Netherlands (4):
  - Radboudumc ( Site 0091), Nijmegen, Gelderland
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 0090), Amsterdam, North Holland
  - Amsterdam UMC, locatie VUmc ( Site 0093), Amsterdam, North Holland
  - Erasmus Medisch Centrum ( Site 0092), Rotterdam, South Holland
- South Korea (4):
  - Seoul National University Hospital ( Site 0150), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0151), Seoul
  - Asan Medical Center ( Site 0153), Seoul
  - Samsung Medical Center ( Site 0152), Seoul
- Spain (4):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 0113), L'Hospitalet de Llobregat, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 0112), Barcelona, Catalonia
  - Hospital Universitario Fundación Jiménez Díaz-START Madrid-FJD ( Site 0111), Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria ( Site 0114), Málaga
- Taiwan (3):
  - Chi Mei Medical Center ( Site 0162), Tainan, Tainan
  - National Cheng Kung University Hospital ( Site 0161), Tainan
  - National Taiwan University Hospital ( Site 0160), Taipei
- Turkey (Türkiye) (4):
  - Ankara Bilkent Şehir Hastanesi. ( Site 0131), Çankaya, Ankara
  - Ankara University Health Practice and Research Hospitals ( Site 0134), Ankara
  - Hacettepe Universite Hastaneleri ( Site 0130), Ankara
  - Koc University, School of Medicine ( Site 0133), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/